CLINICAL TRIAL: NCT03370055
Title: LeucoPatch® in Nonhealing Wounds With Exposed Bone or Tendon Study
Acronym: LiNWEX
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was closed due to lack of participants
Sponsor: Jais Oliver Berg (Other)
Collaborators: Nordsjaellands Hospital (Other); Reapplix (Other)
Responsible Party: Sponsor-Investigator, Jais Oliver Berg, Senior Consultant,, Nordsjaellands Hospital
Organization: Nordsjaellands Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LiNWEX
Record Dates: First submitted 2017-11-20; First posted 2017-12-12 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Wound Healing Delayed
Keywords: Exposed tendon or bone; LeucoPatch; Plastic Surgery; Granulation tissue; Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: observer blinded, randomised, controlled study
Who Masked: Outcomes Assessor
Masking Description: A blinded assessor will evaluate wound healing at the first woundhealing and 2 weeks after woundhealing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LeucoPatch® (Active Comparator): Usual wound care and LeucoPatch® treatment for 8 weeks, with the offer of additional 8 weeks treatment with LeucoPatch®
  Interventions: Device: LeucoPatch®; Other: Control,
- Control (Placebo Comparator): Usual wound care for 8 weeks, with the offer of 8 weeks of LeucoPatch® treatment after the first 8 weeks
  Interventions: Device: LeucoPatch®; Other: Control,

INTERVENTIONS:
Device: LeucoPatch® — LeucoPatch® is an elastic membrane produced by the patients own venous blood by centrifugation, and one or two is placed on the wound once a week The LeucoPatch® consist of the fibrin Leucocytes and growth factors from the patients own blood
Other: Control, — Usual wound care in a specialized clinic

SUMMARY:
The trial compare the healing rate of chronic wounds with exposed tendon or bone ('problematic wound area') with LeucoPatch® treatment for 8 up to 16 weeks in addition to usual care versus usual care.

The healing rate will be measured as relative reduction of 'problematic wound area' at 8 weeks

DETAILED DESCRIPTION:
A certain subpopulation of plastic surgery patients has chronic, non-healing wounds with exposed bone or tendon e.g. located on the scalp or extremities. The chronic non-healing wounds are characterized by no significant wound area reduction within 4 weeks of standard wound treatment. Standard wound treatment includes mechanical or sharp serial debridement and low pressure irrigation for cleansing and wound dressings ensuring moist wound healing. Exposed bone or tendon in a chronic wound can be described as a potentially 'problematic wound area', since the healing by sound granulation tissue from the soft tissue sides of the wound to cover the problematic wound area is often reduced or absent.

The subpopulation is characterized by either referral from other specialties with non-healing wounds of various etiologies and no or limited options of medical, surgical, or reconstructive plastic surgery procedures to treat the wounds; or the wounds are a consequence of previous reconstructive procedures with unsuccessful outcome and no or limited options of further reconstructive surgery. This group of patients often needs wound treatment for a very long period (months-years) to heal, in spite of best practice standards of wound treatment. Treatment with xenogeneic acellular dermal matrixes and autologous full- or split-thickness skin grafts may be an option, but it often requires general anesthesia and a 2-staged approach. The LeucoPatch may be a new solution in wound treatment, which can be used in the outpatient clinic, to promote faster healing in patients with chronic, non-healing wounds with exposed bone or tendon

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained before any trial related procedures are performed
2. Aged ≥18 years
3. A documented clinically relevant history of chronic wound with exposed tendon and/or bone. Chronic is defined as a non-healing wound over the past 4 weeks with standard care in a specialized clinic.
4. 'Problematic wound area' between 0.25 and 10.0 cm2 measured by Image J at S1- irrespective of the total wound size
5. The subject must be willing and able to comply with the trial protocol

Exclusion Criteria:

1. Haemoglobin < 6.0 mmol/l available at screening (see 10.10)
2. Non-compliance with blood-letting
3. Clinically infected wound or suspected osteomyelitis in the wound area
4. For lower extremity wounds: Critical peripheral artery disease (absence of foot pulse and Ankle-Branchial Pressure Index, ABPI <0.9 and ankle blood pressure < 50 mmHg)
5. For lower extremity wounds: History of vascular by-pass graft or other endovascular intervention within 3 months prior to inclusion.
6. Malignancy in the wound area
7. Need for dialysis
8. Hemophilia, leukaemia or other significant blood disease
9. History of alcohol or drug abuse within the last year
10. Weight abnormality (BMI < 20 kg/m2 or >30 kg/m2)
11. Pregnant or lactating woman
12. Women of childbearing potential who are not using sufficient contraceptives
13. Patient has previously been randomised in this study
14. Participation in another investigational drug trial within the last 10 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Healing rate of Problematic wound area | 8 weeks
  Measured as relative reduction of Problematic wound area

SECONDARY OUTCOMES:
Complete 'problematic wound area´coverage | 8 weeks or until 16 weeks
  Full coverage with granulation tissue of the 'Problematic wound area´ making split -thickness-skin-transplantation for full wound coverage possible
Complete healing of target wound | 8 or until 16 weeks
  Defined as confirmed confirmed wound closure of target wound i.e. skin reepithelization without drainage or dressing requirements (sustained for 2 weeks)
Time to complete healing or coverage with granulation tissue | until 16 weeks
  Defined as time from randomisation to first study visit with confirmed healing or coverage with granulation tissue
Long -term followup | 36 weeks
  Occurence of complete healing 36 weeks after randomisation
Local pain | 8 to 16 weeks
  Local pain measured with Visual Analogue Scale (VAS )
Safety | 16 weeks
  Data on adverse events and serious adverse events including major clinical events will be compared between treatment groups as will changes in haemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Lise Tarnow, Professor, Study Chair — Nordsjaellands Hospital
Locations (1):
- Herlev - Gentofte Hospital, Herlev, Regionh, Denmark

IPD SHARING:
Plan to Share IPD: No